CLINICAL TRIAL: NCT03217708
Title: Post Discharge Circadian Dysrhythmias, Sleep Disturbances, and Return to Baseline Activity in Children With Pre-existing Obstructive Sleep Apnea After AT (Adenotonsillectomy).
Brief Title: Post Discharge Circadian Rhythms Post Adenotonsillectomy
Status: Withdrawn | Type: Observational
Why Stopped: Non compliance from sponsor regarding applicable documentation to proceed with trial, therefore decision to permanently halt trial
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Arvind Chandrakantan, Assistant Professor of Anesthesiology and Pediatrics, Baylor College of Medicine
Other Study IDs: H-39906
Record Dates: First submitted 2017-04-25; First posted 2017-07-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Circadian Dysrhythmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Children without OSA: Children for AT due to chronic tonsillitis without OSA.
  Interventions: Device: Jawbone UP4
- Children with OSA: Children with OSA for AT as determined by PSG
  Interventions: Device: Jawbone UP4

INTERVENTIONS:
Device: Jawbone UP4 — Wrist worn wearable technology will be utilized to study HR, temperature, sleep, activity changes before and after surgery.

SUMMARY:
The purpose of this study is to utilize non-invasive, easily measurable biomarkers (heart rate, skin temperature, sleep, and activity) in the post surgical discharge period to identify trends which correlate with improved outcome and early recovery (return to baseline activity). These are measured (captured) utilizing a wearable technology (WT) device.

Return to baseline (RTB) activity for the purpose of this study is defined primarily as step count normalization as a surrogate of activity (pre versus post operative step count), and heart rate variability normalization back to preoperative baseline. Increased heart rate variability has been studied in acute care settings as a marker of poor prognosis. Please note that return to baseline is not defined for the pediatric population in the same way as adults (which is primarily questionnaire based and not applicable in children).

DETAILED DESCRIPTION:
Wearable technology has tremendous advantages over current methods of assessing RTB activity in the post-discharge pediatric population after AT, which rely on quality of life (QOL) scales, caregiver and patient reports, as well as nurse phone calls and office visits. These methods are biased, time and labor intensive, disease focused, and caregiver dependent. The investigators propose to use wearable technology in order to assess RTB activity. The device has validated methodology in sleep metrics (as compared to polysomnography), heart rate and activity monitoring (optical sensor and 3 plane accelerometry), and temperature measuring (galvanic skin resistance). So far, no investigators have utilized wearable technology and biomarker (heart rate, skin temperature, activity, sleep) data in the manner proposed. RTB is a difficult to measure entity in children and the investigators have defined it using step count as a marker of activity. There are no studies or "standard" to measure quality of recovery in children.

ELIGIBILITY:
Inclusion Criteria:

* As stated previously, OSA v. non OSA

Exclusion Criteria:

-

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We are testing variability in circadian biomarkers
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Change in circadian rhythm | 3 week
  HR (heart rate) in OSA (obstructive sleep apnea) group v. non OSA group post AT
Change in circadian rhythm | 3 weeks
  Sleep in OSA group v. non OSA group post AT. Specifically the design will capture sleep metrics (REM v. non REM, arousals, movement) in order to assess sleep quality.
Change in activity | 3 week
  Activity change in OSA group v. non OSA group post AT. Due to the device being able to measure activity (specifically measured as step count as indicated in the introduction), these can be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No